CLINICAL TRIAL: NCT05087264
Title: Single Center Clinical Study of Intravenous Indocyanine Green in Pelvic Nerve Visualization During Radical Hysterectomy for Cervical Cancer
Brief Title: Clinical Study of Indocyanine Green Displaying Pelvic Nerve in Radical Operation of Cervical Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.FK.001
Record Dates: First submitted 2021-09-25; First posted 2021-10-21 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2021-09

CONDITIONS: Cervical Carcinoma
Keywords: Cervical Carcinoma; Indocyanine green; Neural phenomenon; Infrared imaging
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Experimental group, control group
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Indocyanine green injection (Experimental): 43 cases received preoperative intravenous injection of indocyanine green and radical resection of q-mc1 cervical cancer under pelvic autonomic nerve fluorescence development
  Interventions: Drug: Indocyanine green
- Not Indocyanine green injection (No Intervention): 43 cases underwent routine surgery，not indocyanine green injection

INTERVENTIONS:
Drug: Indocyanine green — ICG retention test and clearance test: intravenous injection, 0.5mg/l. Liver blood flow measurement: intravenous drip, dissolve 25mg ICG in 100ml injection water, and drip at a constant speed for about 50min to make the ICG concentration reach equilibrium.
  Arms: Indocyanine green injection

SUMMARY:
Indocyanine green was injected intravenously into patients with cervical cancer before operation. The nerve development was observed by infrared imaging system during operation, which was used as the basis for nerve preserving operation of type C cervical cancer. The recovery of bladder function was observed.

DETAILED DESCRIPTION:
This study is an open, randomized and prospective clinical study. 86 patients are planned to be randomly assigned according to 1:1. 43 patients underwent preoperative intravenous injection of indocyanine green, radical resection of q-mc1 cervical cancer under pelvic autonomic nerve fluorescence, and 43 patients underwent routine surgery to observe the medium and long-term urinary system function and pelvic floor function of the subjects.

Before operation, confirm the pathological type, pelvic and abdominal enhancement CT or MRI examination, urography (if necessary), two researchers with senior professional title of gynecology respectively carry out gynecological double diagnosis and triple diagnosis examination, and carry out clinical staging according to figo2018 staging standard; According to NCCN guidelines, subjects who are suitable for radical resection of q-m type C1 cervical cancer (IB1 stage deep interstitial Infiltrator / ib2-iia2 stage) are enrolled for routine preoperative examination, and surgical contraindications are excluded. The operation method is open radical resection of q-m C1 cervical cancer. The same group of researchers with rich experience in gynecological tumor operation act as the chief surgeon. Gradually open the retroperitoneum, walk along the ureter to complete anatomical exposure, observe and record the fluorescence staining degree of pelvic autonomic nerve at different time nodes, and compare with the surrounding blood vessels / lymphatic vessels / adipose tissue, Observe the bladder branch of pelvic visceral nerve, dissociate the pelvic visceral nerve plexus from the rectum uterus / rectocervical ligament, preserve the nerve tissue behind the ureter and bladder, and perform extensive resection.

The shape map of pelvic autonomic nerve (including near-infrared region I and region II) was developed. The researchers recorded the identification of nerve after operation and recorded the best observation time point.

The researchers recorded the operation time, the amount of bleeding, the length of the resected uterosacral ligament, main ligament and bladder cervical ligament, and the distal margin was reserved for nerve staining and quantitative analysis.

Safety observation: allergic reaction, influence on liver and kidney function, influence on hemagglutination state.

Observation of recent indicators of bladder dysfunction after operation: the catheter was removed 1 week after operation, and the residual urine volume was measured by ultrasonography. The catheter was placed again if it was > 100ml, and then rechecked once a week until the residual urine volume was less than 30ml.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects have certain reading ability, can communicate effectively with the researchers, and voluntarily sign the informed consent form
2. they are 18-75 years old (including the boundary value) and the ECoG score is 0-1
3. Patients with newly diagnosed cervical squamous epithelial carcinoma and cervical adenocarcinoma confirmed by histology
4. according to NCCN guidelines, they are suitable for patients undergoing radical resection of q-m C1 cervical cancer, i.e. IB1 stage deep interstitial infiltrators / ib2-iia2 stage and early IIB stage
5. normal range of liver and kidney function: bilirubin ≤ 1.5 times ULN, ALT and AST ≤ 2.5 times ULN, creatinine ≤ 1.5 times ULN, Or creatinine clearance rate ≥ 50ml / min (using standard Cockroft Gault formula)
6. have good review and follow-up conditions, and be followed up for at least 1 year

Exclusion Criteria:

1. The preoperative clinical stage was unclear and the surgical indications were controversial
2. Previous history of malignant tumor or radiotherapy or chemotherapy or antiangiogenic therapy
3. pathological types are neuroendocrine carcinoma, small cell tumor, clear cell carcinoma, sarcoma and other histological types
4. urinary disease obstruction and hydronephrosis
5. severe congestive heart failure of grade II or above of New York Heart Association, History of myocardial infarction or unstable angina pectoris within 6 months before operation; Stroke or transient ischemic attack within 6 months before operation
6. pregnancy or lactation
7. according to the judgment of the investigator, it may increase the risk related to the study, may interfere with the interpretation of the study results, or the investigator believes that the patients are not suitable for inclusion

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-03-10 (Estimated); Primary Completion 2025-10-16 (Estimated); Study Completion 2025-10-16 (Estimated)

PRIMARY OUTCOMES:
Main indicators of bladder function recovery | 7 days after operation
  Residual urine volume of bladder 7 days after operation

SECONDARY OUTCOMES:
Other indicators of bladder function recovery | 12, 24 and 48 weeks after operation
  ① Micturition time, micturition times, tension urinary incontinence, prolonged micturition time, abdominal pressure micturition, incomplete micturition and dysuria; ② Urodynamic examination, monitoring the maximum urinary flow rate (MFR), average urinary flow rate (AFR), residual urine volume (RU), initial urinary bladder volume (FVS), maximum urinary bladder volume (MVS), detrusor contraction and maximum detrusor contraction force (MDP); ③ Pelvic floor function evaluation: pelvic floor function examination was performed 24 weeks after operation.

CONTACTS AND LOCATIONS:
Locations (1):
- FifthSunYetSen, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No